CLINICAL TRIAL: NCT00466024
Title: Particulate Reduction Education in City Homes (PREACH)
Brief Title: Particulate Reduction Education in City Homes
Acronym: PREACH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Arlene M. Butz, Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 001673; P01 R826724
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Asthma; persistent; children; particulates; ETS
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Health coach and 2 HEPA air cleaners
  Interventions: Behavioral: Health Coach and HEPA Air cleaners
- 2 (Active Comparator): Standard asthma education and 2 HEPA air cleaners
  Interventions: Behavioral: Health Coach and HEPA air cleaners
- 3 (Active Comparator): Standard asthma education and delayed receipt of 2 HEPA air cleaners
  Interventions: Behavioral: Health Coach and HEPA air cleaners

INTERVENTIONS:
Behavioral: Health Coach and HEPA Air cleaners — Health Coach for ETS reduction in home and 2 HEPA air cleaners
  Other Names: Behavior and HEPA
  Arms: 1
Behavioral: Health Coach and HEPA air cleaners — Behavioral training and 2 HEPA air cleaners
  Other Names: Behavior and HEPA

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial of the efficacy of a combination of HEPA room air cleaners plus an ETS reduction behavior training as compared to either HEPA air cleaners plus standard asthma education or delayed HEPA air cleaners and standard asthma education (control group).

DETAILED DESCRIPTION:
150 children aged 6-12 years who reside in Baltimore and have a smoker in the household are to be enrolled in this study. All children will be randomized into three groups: HEPA air cleaners plus ETS/Indoor particulate behavior management, HEPA air cleaners and a standard asthma education and a standard asthma education group with delayed HEPA filter use. The HEPA air cleaner plus ETS/Indoor particulate behavior management intervention group will receive four home visits by a health coach to assess motivation for parental behavior change and then assist the parent to reduce/eliminate their child's exposure to ETS in the home. The intervention is based on the social cognitive theory that utilizes behavior modification techniques (e.g., modeling, reinforcement, self-monitoring, feedback and rehearsal) to change health behaviors. Families in this group and the HEPA air cleaner only group will receive two HEPA air cleaners to use over the 6-month follow-up period and three home visits for standard asthma education. Use of air cleaners will be electronically monitored to determine level or "dose" of air cleaning used by families. The standard asthma education group (delayed HEPA Filter group) will receive three home visits to deliver basic asthma education. All children receive a baseline home inspection, 7-day home PM exposure monitoring, home dust allergen collection, skin testing, urine cotinine, spirometry, serum eosinophilia and exhaled NO testing. Caregivers of each child will be interviewed at baseline and at the 6-month follow-up regarding ETS reduction behaviors in the home, symptom frequency, asthma control, other environmental exposures and health care utilization outcomes. The primary outcome for this study is reduction in PM10 and PM2.5 over the 6 month follow-up. Secondary outcomes include ETS reduction behavior change (i.e. smoker is smoking outside of home, child not sitting with smoker, reduction in number of household smokers), symptom free days and health care utilization measures. If successful, this intervention could have significant clinical and public health applications for pediatric asthma management in children with persistent asthma and high ETS home exposure.

ELIGIBILITY:
Inclusion Criteria:

* An eligible child will be defined as:

  * Age 6-12 years
  * Doctor's diagnosis of asthma
  * Currently having persistent asthma, defined as asthma symptoms or use of quick reliever asthma medication > 2 days/week in the last 2 weeks or use of daily controller asthma medication in past 2 weeks based on parent report.
  * Reside in eligible household at least 5 days per week

Household:

* Located in Baltimore
* Housing an eligible child
* Housing an English speaking family
* Housing at least one smoker, who smokes 5 or more cigarettes per day. Smoking in the car will be recorded, but if ETS exposure is limited to the car, the household is not eligible.
* Having working electricity and no major structural damage.
* Having no working air cleaner

Exclusion Criteria:

* Children will be excluded is they have other respiratory morbidity such as cystic fibrosis or bronchopulmonary dysplasia, if they smoke cigarettes, if they do not have asthma symptoms or medication use in the month before randomization
* Families living in a shelter or transitional housing will be excluded

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2006-10; Primary Completion 2009-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome for this study is reduction in PM10 and PM2.5 over the 6 month follow-up. | 6 months

SECONDARY OUTCOMES:
Secondary outcomes include ETS reduction behavior change (i.e. smoker is smoking outside of home, child not sitting with smoker, reduction in number of household smokers), symptom free days and health care utilization measures. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Arlene M Butz, ScD, RN, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Butz AM, Matsui EC, Breysse P, Curtin-Brosnan J, Eggleston P, Diette G, Williams D, Yuan J, Bernert JT, Rand C. A randomized trial of air cleaners and a health coach to improve indoor air quality for inner-city children with asthma and secondhand smoke exposure. Arch Pediatr Adolesc Med. 2011 Aug;165(8):741-8. doi: 10.1001/archpediatrics.2011.111. PMID 21810636